CLINICAL TRIAL: NCT01051297
Title: Patients With Obstructive Sleep Apnea (OSA), Independent of Obesity, Are at Increased Risk of Venous Thromboembolic Events (VTE)
Brief Title: Obstructive Sleep Apnea and Venous Thromboembolism
Acronym: OSAVTE
Status: Terminated | Type: Observational
Why Stopped: Investigator left the institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1132357
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Obstructive Sleep Apnea; Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism
Keywords: Obstructive sleep apnea; venous thrombosis; pulmonary embolism; venous thromboembolism
MeSH Terms: conditions — Sleep Apnea, Obstructive; Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- VTE -PROSPECTIVE: Patients diagnosed with VTE
- sleep study group -PROSPECTIVE: patients undergoing sleep study
- VTE-Retrospective: patients with VTE , chart review
- OSA-retrospective: PATIENT WITH OSA -CHART REVIEW
- OSA group -PROSPECTIVE: patients diagnosed with OSA

SUMMARY:
There is a clear link between obstructive sleep apnea (OSA) and cardiovascular disease. However, there has been no clear link between OSA and venous thromboembolism (VTE). The objective of this study is to evaluate such a link.

DETAILED DESCRIPTION:
Design:

1. retrospective chart review of all patients with VTE over 10 year period
2. retrospective chart review of all patients with OSA over 10 year period
3. prospective 1 year follow up of all patients diagnosed with new VTE
4. prospective 1 year follow up of all patients undergoing sleep study

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years) with sleep study, OSA or VTE

Exclusion Criteria:

* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>=18 years) with sleep study , OSA or VTE
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2009-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
incidence of VTE for the OSA cohort | 12 months
incidence of OSA for the VTE cohort | 12 months

SECONDARY OUTCOMES:
death | 12 month
bleeding | 12 months
composite outcome of death, VTE , or bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: OUSAMA DABBAGH, MD, Principal Investigator — University of Missouri-Columbia; JAMES P BOSANQUET, MD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosanquet JP, Bade BC, Zia MF, Karo A, Hassan O, Hess BT, Dabbagh O. Patients with venous thromboembolism appear to have higher prevalence of obstructive sleep apnea than the general population. Clin Appl Thromb Hemost. 2011 Nov-Dec;17(6):E119-24. doi: 10.1177/1076029610389023. Epub 2010 Dec 15. PMID 21159707